CLINICAL TRIAL: NCT00879957
Title: Comparison of Heparin vs. no Heparin on Duration of Peripherally Inserted Central Catheter Patency in Neonates
Brief Title: Heparin Versus no Heparin on Duration of Peripherally Inserted Central Catheter (PICC) Patency in Neonates
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: A study was published regarding the same question this study had.
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Aaron Reeves, MD, University of Texas Health Science Center at San Antonio
Allocation: Non-Randomized | Model: Single Group | Masking: Triple | Purpose: Prevention
Other Study IDs: HSC20090136H
Record Dates: First submitted 2009-03-26; First posted 2009-04-13 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-04

CONDITIONS: Infant, Premature; Anticoagulants; Thrombosis
Keywords: Infant, Premature; Infant; Central venous catheterization; Anticoagulants
MeSH Terms: conditions — Premature Birth; Thrombosis | interventions — Heparin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Heparin group (Active Comparator): The heparin group is the arm of the study in which all of the subjects will be treated according to current standard medical therapy. All fluids to be infused through their PICCs will have 0.5 units heparin per milliliter of intravenous fluid.
  Interventions: Drug: heparin
- No heparin group (Experimental): This group will only receive the prescribed fluids to infuse through their PICCs. No heparin will be added to the intravenous infusions.
  Interventions: Drug: No heparin

INTERVENTIONS:
Drug: heparin — Heparin will be added to PICC infusions at a dose of 0.5 units heparin per milliliter of intravenous fluid/parenteral nutrition.
  Arms: Heparin group
Drug: No heparin — In the no heparin group, the subjects will not receive heparin as an additive to their PICC infusions.
  Arms: No heparin group

SUMMARY:
Background: Heparin is an anticoagulant commonly used in the neonatal population as a means to prevent catheter related occlusion and malfunction by thrombosis (clot). Given the recent overdoses of infants using heparin, there is concern as to whether heparin should be used in peripherally inserted central venous catheters (PICC). Scientific evidence comparing the duration of use of heparin versus no heparin in PICCs is conflicting.

Purpose: The purpose of this study is to evaluate the effect of continuous IV fluids with heparin versus IV fluids without heparin on the duration of percutaneously inserted central venous catheters (PICC) in neonates.

Design: Prospective, double-blind, randomized controlled trial Hypothesis: The use of heparin in PICC fluids has no difference on duration of catheter patency.

Design and Methods: The study will be conducted at the Neonatal Intensive Care Unit at University Hospital, San Antonio, TX. Randomization to either the experimental group (no-heparin) or the standard medical group (with heparin) will occur once parental consent is obtained and prior to PICC insertion. PICC placement will be done by the PICC certified neonatal nurses. Correct placement of the PICC will be assured by radiography which is standard procedure.

Parents, NICU team members and staff, and investigators will be masked to the grouping. Pharmacy will be responsible for randomization. Both the heparin group and the no heparin group solutions will be dispensed in identical containers, compounded by the pharmacy.

The study medication, heparin, will be mixed by the pharmacy at a standard dose of 0.5 units/mL for the intravenous infusions used in the heparin group. The experimental group will receive only the base solution, whether it is 5% dextrose, 0.9% sodium chloride, or total parenteral nutrition infused into the PICC line. Pharmacy and the NICU staff will ensure compatibility of heparin with other infusions. Heparin bonded catheters, heparin flushes, and hep-lock solutions are not used by the NICU service.

The primary outcome, duration of catheter use, is defined as the time (in hours) between insertion and removal of the catheter due to occlusion. Occlusion will be defined as the inability to push 1 mL of 0.9% sodium chloride, via a 5 mL syringe, through the catheter in situ or detection of clots along the catheter after removal.

Secondary outcomes include septicemia vs. catheter-related septicemia, phlebitis, death before discharge, and thrombosis. Septicemia is identified as clinical signs and symptoms associated with sepsis in the presence of a positive peripheral blood culture obtained irrespective of the catheter tip culture result. Catheter-related sepsis will be defined as positive blood culture obtained from the catheter fluid as well as a positive blood culture obtained from a peripheral venous specimen. Both cultures must demonstrate the same organism. Phlebitis is defined by visual detection, swelling, and change of skin color associated with an inflamed vein. Thrombosis is defined as a thrombus along catheter path diagnosed by visual inspection upon removal of the catheter. Elective versus non-elective removal will also be recorded.

Adverse events monitored include: heparin induced thrombocytopenia (HIT), defined as a platelet count dropping below 50 x 103/mL with a positive antibody titer, aPTT > 100 seconds (This will be measured upon clinical evidence of bleeding), hemorrhage from > 2 sites, intraventricular hemorrhage, extravasation, and dislodgement or breakage of catheter.

The sample size will be determined based on retrospective data collection to reach a statistical power of 80% with a type I error or 0.05. The investigators expect the sample size to be approximately 102 patients in each arm of the study.

The study will terminate once the PICC is discontinued or if there is an indication to stop the study early for safety reasons. These could include increased adverse events in one group versus the other. A Safety Control Panel composed of 2 neonatologists from another site will review the data at the points when 1/3 and then 2/3 of total patient enrollment has been achieved.

Data Collection and Analysis: Data will be collected and tabulated on a Microsoft Excel spreadsheet using unique patient identifiers and stored at a secure location at UHS then analyzed using appropriate statistical tests.

ELIGIBILITY:
Inclusion Criteria:

* Neonates admitted to the Neonatal Intensive Care Unit (NICU) at University Hospital in San Antonio, Texas who require a percutaneous central venous catheter, as determined by the attending neonatologist.

Exclusion Criteria:

* Evidence of bleeding (prolonged aPTT)
* Recent sepsis (w/in 48 hours of initiation of antimicrobial therapy)
* Propensity for stroke or thrombophilia
* Requiring heparinization (i.e. dialysis)
* Discretion of the neonatologist (severe illness to the point of uncertain viability, poor intravenous access requiring surgical placement of a long term intravenous catheter e.g. Broviac)
* Requirement of a 1 French catheter
* Uncertain viability (this is based on the discretion of the infant's neonatologist who is not a member of the research team)
* Nonviable neonates (this is based on the discretion of the infant's neonatologist who is not a member of the research team)

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2010-01; Primary Completion 2011-03 (Estimated); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be duration of catheter patency, as defined by the length of time between insertion and removal of the PICC due to catheter occlusion. | 1 day to 3 months

SECONDARY OUTCOMES:
Bacteremia | 1 day to 3 months
Catheter-related bacteremia | 1 day to 3 months
Phlebitis | 1 day to 3 months
Thrombosis | 1 day to 3 months
Death | 1 day to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Aaron A Reeves, M.D., Principal Investigator — The University of Texas Health Science Center at San Antonio; Cynthia L Blanco, M.D., Study Director — The University of Texas Health Science Center at San Antonio
Locations (1):
- University Hospital, San Antonio, Texas, United States

REFERENCES:
- [Background] Moclair A, Bates I. The efficacy of heparin in maintaining peripheral infusions in neonates. Eur J Pediatr. 1995 Jul;154(7):567-70. doi: 10.1007/BF02074836. PMID 7556325
- [Background] Klenner AF, Fusch C, Rakow A, Kadow I, Beyersdorff E, Eichler P, Wander K, Lietz T, Greinacher A. Benefit and risk of heparin for maintaining peripheral venous catheters in neonates: a placebo-controlled trial. J Pediatr. 2003 Dec;143(6):741-5. doi: 10.1016/j.jpeds.2003.09.024. PMID 14657819
- [Background] Shah PS, Kalyn A, Satodia P, Dunn MS, Parvez B, Daneman A, Salem S, Glanc P, Ohlsson A, Shah V. A randomized, controlled trial of heparin versus placebo infusion to prolong the usability of peripherally placed percutaneous central venous catheters (PCVCs) in neonates: the HIP (Heparin Infusion for PCVC) study. Pediatrics. 2007 Jan;119(1):e284-91. doi: 10.1542/peds.2006-0529. PMID 17200252
- [Background] Kamala F, Boo NY, Cheah FC, Birinder K. Randomized controlled trial of heparin for prevention of blockage of peripherally inserted central catheters in neonates. Acta Paediatr. 2002;91(12):1350-6. doi: 10.1111/j.1651-2227.2002.tb02833.x. PMID 12578294
- [Background] Shah PS, Shah VS. Continuous heparin infusion to prevent thrombosis and catheter occlusion in neonates with peripherally placed percutaneous central venous catheters. Cochrane Database Syst Rev. 2008 Apr 16;2008(2):CD002772. doi: 10.1002/14651858.CD002772.pub3. PMID 18425882
- [Background] de Neef M, Heijboer H, van Woensel JB, de Haan RJ. The efficacy of heparinization in prolonging patency of arterial and central venous catheters in children: a randomized double-blind trial. Pediatr Hematol Oncol. 2002 Dec;19(8):553-60. doi: 10.1080/08880010290097404. PMID 12487830